CLINICAL TRIAL: NCT06805903
Title: Adherence Assessment in Transanal Irrigation : Validation of the Transanal Irrigation Adherence Scale
Brief Title: Validation of TRansanal Irrigation Adherence scaLe (TRIAL)
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP241770
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Irritation; Anus
Keywords: transanal irrigation; adherence; bowel dysfonction; constipation; fecal incontinence
MeSH Terms: conditions — Constipation; Fecal Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: TRansanal Irrigation Adherence scaLe — new trans-anal irrigation self-assessment questionnaire in French

SUMMARY:
Transanal irrigation (TAI) is a method used to empty stools from the recto-sigmoid and colon (from the descending colon to the transverse colon). It is recommended for treating evacuation disorders (bowel movements) or continence issues (fecal incontinence). It is a second-line treatment, offered after the failure of hygienic-dietary rules, perineal physiotherapy, and conventional drug treatments (suppositories, obturator plugs, etc.), in combination with treatments for transit constipation (hygienic-dietary rules and laxatives) if necessary.

The effectiveness of TAI has been widely demonstrated, particularly in neurological populations (spinal cord injuries, spina bifida, multiple sclerosis, etc.), but also in non-neurological populations, with a significant reduction in symptoms (constipation or incontinence) and an improvement in quality of life compared to medical treatment Despite demonstrated effectiveness with a long-term success rate of 50% among users, only 42% of patients continue use 21 months after learning the technique.

The aim of this study is to validate a tool for assessing patient adherence to the TAI device in order to identify non-adherent patients and subsequently determine the reasons for non-adherence to optimize treatment, in the absence of non-surgical therapeutic alternatives The primary objective of this study is the psychometric validation of a transanal irrigation adherence self-questionnaire scale (TRIAL) in French.

The secondary objectives are assessing : 1/ correlation between the final score of TRIAL with sides effects reported, the using modalities, indications of this treatment, and patient's satisfaction. 2/ quality of life of these patients using the Transanal irrigation device. 3/ correlation between the final score of TRIAL and stool diary in order to define the cut-offs of strong, moderate and low adherence of this scale.

DETAILED DESCRIPTION:
Transanal irrigation (TAI) is a method used to empty stools from the recto-sigmoid and colon (from the descending colon to the transverse colon). It is recommended for treating evacuation disorders (bowel movements) or continence issues (fecal incontinence). It is a second-line treatment, offered after the failure of hygienic-dietary rules, perineal physiotherapy, and conventional drug treatments (suppositories, obturator plugs, etc.), in combination with treatments for transit constipation (hygienic-dietary rules and laxatives) if necessary.

The effectiveness of TAI has been widely demonstrated, particularly in neurological populations (spinal cord injuries, spina bifida, multiple sclerosis, etc.), but also in non-neurological populations, with a significant reduction in symptoms (constipation or incontinence) and an improvement in quality of life compared to medical treatment Despite demonstrated effectiveness with a long-term success rate of 50% among users, only 42% of patients continue use 21 months after learning the technique.

The aim of this study is to validate a tool for assessing patient adherence to the TAI device in order to identify non-adherent patients and subsequently determine the reasons for non-adherence to optimize treatment, in the absence of non-surgical therapeutic alternatives

The primary objective of this study is the psychometric validation of a transanal irrigation adherence self-questionnaire scale (TRIAL) in French.

The secondary objectives are assessing : 1/ correlation between the final score of TRIAL with sides effects reported, the using modalities, indications of this treatment, and patient's satisfaction. 2/ quality of life of these patients using the Transanal irrigation device. 3/ correlation between the final score of TRIAL and stool diary in order to define the cut-offs of strong, moderate and low adherence of this scale.

Inclusions will be headed during a consultation or a one day follow-up hospitalization in a neuro-urology department. On this day, patients will have a medical consultation and data concerning medical history, treatments, pelvic disorders' characteristics and modalities of use of TAI will be recorded. The patient will also complete the following questionnaires: TRIAL, a numeric scale of TACI effectiveness, Kess, Wexner, STAR-Q (if diagnosed with multiple sclerosis), NBD (if spinal cord injury), which are symptom scores for ano-rectal disorders; PGI-Severity of ano-rectal disorders; PGI-Improvement of ano-rectal disorders with TACI; USP; I-CAS (if using self-catheterization); and a numeric scale assessing the impact of ano-rectal disorders on quality of life.

Then, at home, the patient will complete a diary detailing the frequency of TAI use over 15 days, along with a new TRIAL questionnaire on day 15, which will be mailed back using a pre-stamped envelope provided by the department.

The validation of this new scale about TAI's adherence is part of a will to standardize the evaluation especially in the use of this device in order to identify the difficulties encountered by patients within therapeutic education programs for learning this technique.

ELIGIBILITY:
Inclusion criteria

* Patients using ICT for at least 1 month
* Patients with anorectal disorders of neurological or neurological or non-neurological origin
* Patients whose indication for TCI is constipation, anorectal and/or fecal incontinence.
* Adult patients
* Informed patients who do not object to participating in the study.

Exclusion criteria

* Language barrier and comprehension difficulties
* Patients under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women over 18 years old using transanal irrigation device
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Psychometric validation of a transanal irrigation adherence self-questionnaire scale, in French | 30 months and 15 days

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.